CLINICAL TRIAL: NCT04965506
Title: A Randomized Phase II Study to Evaluate the Efficacy and Safety of IBI362 Versus Placebo and Dulaglutide in Chinese Patients With Type 2 Diabetes
Brief Title: A Study of IBI362 in Chinese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362A201
Record Dates: First submitted 2021-07-15; First posted 2021-07-16 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mazdutide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IBI362 low dose (Experimental): Participants receive low dose IBI362 by subcutaneous (SC) injection once a week.
  Interventions: Drug: IBI362
- IBI362 moderate dose (Experimental): Participants receive medium dose IBI362 by subcutaneous (SC) injection once a week.
  Interventions: Drug: IBI362
- Dulaglutide (Active Comparator): Participants receive Dulaglutide 1.5mg by subcutaneous (SC) injection once a week.
  Interventions: Other: Dulaglutide
- IBI362 high dose (Experimental): Participants receive high dose IBI362 by subcutaneous (SC) injection once a week.
  Interventions: Drug: IBI362
- placebo (Placebo Comparator): Participants receive placebo by subcutaneous (SC) injection once a week.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: IBI362 — IBI362 administered subcutaneously (SC) once a week.
  Arms: IBI362 high dose; IBI362 low dose; IBI362 moderate dose
Other: placebo — placebo administered subcutaneously (SC) once a week.
  Arms: placebo
Other: Dulaglutide — Dulaglutide administered subcutaneously (SC) once a week.
  Arms: Dulaglutide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IBI362 in Chinese patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Have type 2 diabetes (T2DM) for ≥6 months according to the Criteria for Diagnosing Type 2 Diabetes Mellitus (WHO 1999)
2. T2D patients with poorly controlled blood glucose treated with lifestyle intervention or stable dose of metformin (≥ 1000mg/day or maximum tolerated dose) within 3 months prior to screening.
3. Have HbA1c of 7.0% to 10.5%, inclusive(detected by local laboratory at screening).
4. Have a body mass index (BMI) between 20(Inclusive) and 40 kilograms per square meter

Exclusion Criteria:

1. Type 1 diabetes, special types of diabetes, or gestational diabetes.
2. Have uncontrolled diabetes defined as more than 2 episodes of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to screening.
3. History of severe hypoglycemic episodes within 6 months prior to screening.
4. Have had any of the following within the last 6 months prior to screening: myocardial infarction (MI), unstable angina, coronary artery bypass graft, percutaneous coronary intervention (diagnostic angiograms are permitted),transient ischemic attack (TIA), cerebrovascular accident or decompensated congestive heart failure, or currently have New York Health Association Class III or IV heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
The change in HbA1c from baseline to 20 weeks | Baseline,20 weeks

SECONDARY OUTCOMES:
Percentage of Participants Achieving HbA1c Target of <7.0% | Baseline,20 weeks
Number of participants with treatment-related adverse events | Baseline,25 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No